CLINICAL TRIAL: NCT00344851
Title: Comparison of the Effects of Monotherapy With Exenatide or Metformin to Combined Exenatide and Metformin Therapy on Menstrual Cyclicity in Overweight Women With Polycystic Ovary Syndrome
Brief Title: Exenatide and Metformin Therapy in Overweight Women With PCOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metabolic Center of Louisiana Research Foundation (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP06-010
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2007-07-11 (Estimated); Status verified 2007-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: menstrual cyclicity; insulin resistance; body fat distribution; pancreatic ß-cell function; inflammatory markers; liver function tests
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: metformin, exenatide or combined (metformin & exenatide )

SUMMARY:
Current research has shown that the use of diabetes management practices aimed at reducing insulin resistance and hyperinsulinemia (such as weight reduction and the administration of oral antidiabetic drugs) in women with PCOS can not only improve glucose and lipid metabolism but can also reverse testosterone abnormalities and restore menstrual cycles. A new medicine called exenatide (Byetta) has been found to reduce body weight, as well as, improve abnormal glucose metabolism in diabetics. This randomized study will compare Exenatide (Byetta) to extended release metformin (Fortamet) to combination therapy (both Byetta and Fortamet) on menstrual cyclicity, hormone profiles and metabolic profiles over a 24-week period in women with PCOS.

DETAILED DESCRIPTION:
Objectives: The objective of the present proposal is to compare the clinical, endocrine and metabolic effects of therapy with exenatide and metformin alone, to combination therapy in women with PCOS. This study will serve as a pilot investigation to open perspectives for future investigations combining insulin-sensitizing drugs with different mechanisms of action in patients with PCOS, especially ones for whom standard treatment with metformin is less effective.

Subjects : 60 oligomenorrheic overweight/obese (BMI >27) women meeting criteria for PCOS (age 18-40)· six or fewer menses /year or amenorrheic· clinical or laboratory evidence of hyperandrogenism (hirsutism or elevated testosterone (T))· PCOS ovary on ultrasound(need to meet criteria 1 and either 2 or 3 [or both]) Inclusion/Exclusion Criteria: Major EXCLUSION CRITERIA - FEMALE1) other uncorrected endocrinopathy- hyperprolactinemia, hyper- or hypothyroidism, congenital adrenal hyperplasia2) presence of overt diabetes or impaired glucose tolerance3) alterations in hepatic or renal function4) use of hormonal medications, insulin sensitizers or medications that interfere with carbohydrate metabolism for at least 8 weeks5) Any medical condition which, in the judgment of the investigator may interfere with the absorption, distribution, metabolism or excretion of the drug6) Simultaneous participation in another clinical trial7) Known active substance abuse including tobacco and alcohol. (> 10 cigarettes/day)8) Refusal or inability to comply with protocol9) patient desiring pregnancy, pregnant, or breastfeeding Study Design: Balanced randomized parallel group clinical study with 3 treatment arms: metformin (1000 mg BID); exenatide (10 mcg BID) or combined (metformin 1000 mg BID; exenatide 10 mcg BID) therapy for 24 weeks.

Efficacy Measures: Primary- Menstrual Cyclicity ( # menses/ 24 weeks)Secondary-BMI, WHR, FAI (T/SHBG), DHEAS, lipids, insulin resistance-(HOMA and composite insulin sensitivity index [ SIOGTT), and pancreatic ß-cell function (corrected insulin response [CIRgp] and insulinogenic index [IGI] ).

Safety: For safety, all subjects who enter the study are evaluable. Subjects will be monitored for safety by assessment of adverse events, physical exams, vital signs and laboratory values.

Statistical methods/analysis: The measurement of menstrual frequency involves nominal data ( patients with/without regular cycles pre vs post-treatment and will be analyzed using the McNemar test (complex chi square for paired data). For all other analyses, in which the data are interval, parameters, such as androgens, lipids, insulin sensitivity, etc. will be evaluated using a SS/Treatment x Trials (pre/post) analyses of variance (ANOVA). This repeated measures design will allow us to determine if each of the treatment drugs had an effect and if they are significantly different from each other while controlling for individual patient differences Study Drug Regimens: Exenatide5 ug bid - 4 weeks10 ug bid - 20 weeks (end of study)Metformin500 mg qd 2 weeks500 mg bid 2 weeks 500 mg am, 1000 mg pm- 2 weeks1000 mg bid -18 weeks (end study) Exenatide plus MetforminExenatide- 5 ug bid-4 weeksMetformin 500 qd for 2 weeks, 500 mg bid 2 weeksExenatide- 10 ug -20 weeks (to end of study)Metformin-500 mg am, 1000 mg pm- 2 weeks - 1000 bid for 18 weeks (end of study)** Metformin may be adjusted at the discretion of the physician to a level that is tolerable in patients who cannot tolerate the full dose of metformin in combination with exenatide (combination therapy only )

ELIGIBILITY:
Inclusion Criteria:Overweight/obese women (BMI>27)

1. Must have six or fewer menses /year or be amenorrheic
2. Have either clinical or laboratory evidence of hyperandrogenism (hirsutism or elevated testosterone (T)) and /or PCOS ovary on ultrasound

Exclusion Criteria:

other uncorrected endocrinopathy- hyperprolactinemia, hyper- or hypothyroidism, congenital adrenal hyperplasia or presence of overt diabetes alterations in hepatic or renal function use of hormonal medications, insulin sensitizers or medications that interfere with carbohydrate metabolism for at least 8 weeks Known active substance abuse including tobacco and alcohol. Pregnancy, breastfeeding or desire for pregnancy during study interval (6 months

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
- Menstrual Cyclicity ( # menses/ 24 weeks) | every 4 weeks

SECONDARY OUTCOMES:
BMI, WHR, FAI (T/SHBG), DHEAS, lipids,abdominal girth, | BMI,WHR,abdominal girth at start,12 weeks and 24 weeks, FAI, DHEAS, lipids at start and at 24 weeks
insulin resistance-(HOMA and composite insulin sensitivity index [ SIOGTT), | at start and at 24 weeks
and pancreatic ß-cell function (corrected insulin response [CIRgp] and | at start and at 24 weeks
insulinogenic index [IGI] ). | at start and at 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Elkind-Hirsch, Ph.D., Principal Investigator — Woman's Health Research Institute; Rajat Bhushan, M.D., Principal Investigator — Metabolic Center of Louisiana Resarch Foundation
Locations (1):
- Facility: Metabolic Center of Louisiana Research Foundation, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Elkind-Hirsch K, Marrioneaux O, Bhushan M, Vernor D, Bhushan R. Comparison of single and combined treatment with exenatide and metformin on menstrual cyclicity in overweight women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2008 Jul;93(7):2670-8. doi: 10.1210/jc.2008-0115. Epub 2008 May 6. PMID 18460557